CLINICAL TRIAL: NCT00441649
Title: Methylphenidate Treatment of ADHD in Children With Tourette Syndrome
Brief Title: Methylphenidate for Treating Children With ADHD and Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH045358 (NIH); R01MH045358 (NIH); DDTR B2-NDH
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Tourette Syndrome
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Tourette Syndrome | interventions — Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate

SUMMARY:
This study will evaluate the safety and effectiveness of methylphenidate in treating attention deficit hyperactivity disorder in children with both attention deficit hyperactivity disorder and Tourette syndrome.

DETAILED DESCRIPTION:
Tourette syndrome is a neurological disorder that is characterized by repetitive, involuntary movements and vocalizations called tics. Many children with Tourette syndrome also have attention deficit hyperactivity disorder (ADHD), which is one of the most common childhood mental disorders. Symptoms of ADHD usually include impulsiveness, inattention, and hyperactivity. ADHD is commonly treated with a stimulant medication, such as methylphenidate. It is under debate, however, whether using stimulants in children with Tourette syndrome exacerbates tics associated with the disorder. This study will evaluate the safety and effectiveness of methylphenidate in treating ADHD in children who have both ADHD and Tourette syndrome.

Participants in this 6-week, double blind study will receive three doses of methylphenidate over the course of the study. Each dose will be taken twice daily, approximately 3.5 hours apart, for 2 weeks. Medication will be dispensed at study visits, which will occur once every 2 weeks. At each study visit, participants will take a dose of the medication. About an hour after ingesting the medication, they will be observed in a classroom setting by study physicians. Participants will then complete a Continuous Performance Test, which will measure their voluntary attention levels. The following will be assessed at study visits: ADHD symptoms; oppositional and aggressive behavior; frequency and severity of tics and obsessive compulsive disorder symptoms; rebound tic exacerbation; effects of methylphenidate on tic-related problems with self-esteem, family life, academic and social performance, and overall tic severity; anxiety and mood symptoms; and adverse drug reactions. Parents and teachers will also complete assessments of participants' behavior on 2 days of each week for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD or ADHD plus Tourette syndrome

Exclusion Criteria:

* Determined to be dangerous to self or others
* Scores less than 70 on an IQ test
* Any seizure disorder, major organic brain dysfunction, major medical illness, major mood disorder, psychosis, pervasive developmental disorder, or peripheral sensory loss
* Any condition that may make use of methylphenidate unsafe

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71
Dates: Start 2000-02; Primary Completion 2004-06 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
ADHD symptoms
Oppositional and aggressive behavior
Frequency and severity of tics and obsessive compulsive disorder symptoms
Tic impairment, tic severity, and clinical response
Anxiety and mood symptoms
Rebound tic exacerbation
Adverse drug reactions (all measured at 2-week intervals throughout the study)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D. Gadow, PhD, Principal Investigator — State University of New York at Stony Brook

REFERENCES:
- [Background] Gadow KD, Sverd J, Sprafkin J, Nolan EE, Ezor SN. Efficacy of methylphenidate for attention-deficit hyperactivity disorder in children with tic disorder. Arch Gen Psychiatry. 1995 Jun;52(6):444-55. doi: 10.1001/archpsyc.1995.03950180030005. PMID 7771914
- [Background] Gadow KD, Sverd J, Sprafkin J, Nolan EE, Grossman S. Long-term methylphenidate therapy in children with comorbid attention-deficit hyperactivity disorder and chronic multiple tic disorder. Arch Gen Psychiatry. 1999 Apr;56(4):330-6. doi: 10.1001/archpsyc.56.4.330. PMID 10197827